CLINICAL TRIAL: NCT03733366
Title: Effects of Different Desktop Materials on Thermal Comfort and Attention
Brief Title: Thermal Comfort of Different Desktop Materials
Acronym: Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: Innorenew CoE (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Thermal comfort
Record Dates: First submitted 2018-10-29; First posted 2018-11-07 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2018-11

CONDITIONS: Office Desk Ergonomics
Keywords: desk surface; thermal comfort; ergonomics; attention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Desk surface — The participants will test all 10 desk surfaces and will be randomly allocated to one of the desks each time.

SUMMARY:
The aim of this study is to test the suitability of different types of desk surfaces. The investigators will test 10 different surfaces (oak-ruff, oak-varnished, oak-oiled, spruce-ruff, spruce-varnished, spruce-oiled, particleboard laminate, particleboard veneer, corian and glass). Firstly, the investigators will perform tests to assess physical characteristics of the materials (thermal conductivity, hardness, roughness, skid measures). Secondly, the investigators will measure the participants' forearm skin temperature after 20-minutes of using each desk surface. During those 20 minutes the participants will solve an attention test.

DETAILED DESCRIPTION:
People are surrounded by objects that are made of different materials. These materials should be carefully chosen, especially the ones that are in direct contact with user's skin. Office workers are constantly in contact with desk surface (while reading, typing, filling in forms, etc.). Therefore, it is important that the material of desk surface is suitable and properly chosen. It should be both functional and aesthetic. The aim of this study is to evaluate the suitability of different desk surfaces for sedentary workers. The investigators will test 10 different surfaces (oak-ruff, oak-varnished, oak-oiled, spruce-ruff, spruce-varnished, spruce-oiled, particleboard laminate, particleboard veneer, corian and glass). All surfaces will be square shaped (800x800 mm). Firstly, the investigators will perform tests to assess physical characteristics of the materials (thermal conductivity, hardness, roughness, skid measures). Secondly, the investigators will measure the participants' forearm skin temperature after 20-minutes of desk use. Every participant will test all 10 sample desk surfaces (cross-over design). The investigators will use thermal IR camera to measure the temperature of participant's skin surface. The investigators will measure the temperature before and after the contact with desk surface. During those 20 minutes the participant will solve an attention test to assess the impact of different materials on attention. At the end, the participants will answer a questionnaire about the suitability of the material.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 35

Exclusion Criteria:

* pregnancy
* pain presence in any musculoskeletal part > 3 on 10-level scale

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change of the skin temperature measured on forearm | at the beginning and after 20 minutes of using desk surface
  Skin temperature in the forearm will be measured with Infrared thermal camera. Thermal camera is suitable for the measurements since it is a reliable tool for measuring skin temperature. The temperature is presented in Celsius degrees. Moreover, thermal camera provides a thermal picture indicating temperature distribution in the space.

SECONDARY OUTCOMES:
Attention test | 180 seconds
  The attention test will be performed on computer. On the computer screen letters P and R will appear. Each time the letter R appears the participant will have to click ''space''. If a letter P appears the participant should not react.
Adjusted Mood and feelings questionnaire | 180 seconds
  The questionnaire consists of two questions. One is asking the participant about their current mood. The second question is asking the participant about their current arousal. The participant answers both questions using a 9-level scale (1 meaning not at all and 9 meaning very much). There is no total value of the questionnaire. Also, higher or lower values do not represent better or worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nejc Sarabon, PhD, Principal Investigator — Faculty of health sciences, University of Primorska
Locations (1):
- Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No